CLINICAL TRIAL: NCT01468220
Title: Normobaric Hypoxic Training Compared to Ambient Training on the Course of the Metabolic Syndrome
Brief Title: Normobaric Hypoxic Training and Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Michael Boschmann, MD, Research Associate, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Hypoxitrain 1; Hypoximet 1 (Other Grant/Funding Number: DFG_LU_435_12/1)
Record Dates: First submitted 2011-09-15; First posted 2011-11-09 (Estimated); Last update posted 2019-03-04 (Actual); Status verified 2019-03

CONDITIONS: Metabolic Syndrome
Keywords: tissue metabolism; skeletal muscle; adipose tissue; HIF
MeSH Terms: conditions — Metabolic Syndrome | interventions — Endurance Training

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- normoxic training (Placebo Comparator): 6 weeks of endurance training under normoxia
  Interventions: Other: Endurance training
- hypoxic training (Active Comparator): 6 weeks of endurance training under hypoxia
  Interventions: Other: Endurance training

INTERVENTIONS:
Other: Endurance training — Endurance training three times per week over six weeks

SUMMARY:
The patient numbers with metabolic syndrome and diabetes have doubled in the last decade. Data that physical exercise ameliorates the metabolic syndrome are convincing, although the mechanisms of the effect in man are not clear. Numerous endocrine or molecular mechanisms modified by physical exercise are known to be hypoxia-sensitive, i.e. by hypoxia-inducible factor-1 (HIF-1) regulation. Thus, relative hypoxia may link physical exercise and modification of endogenous metabolism. Medical communities seem ill equipped to address the primary issues involved. The investigators have experience with normobaric "hypoxia chambers" and will now test a (physical exercise) training program, using state-of-the-art assessments available nowhere else in Germany. The investigators will compare hypoxia chamber, to ambient training, to test the notion that specific exercise conditions could regulate specific molecular pathways involved in the pathogenesis of the metabolic syndrome. Indeed, hypoxia chamber training could be superior to conventional training in terms of reducing cardiovascular risk factors or improving fitness. The investigators will test overall metabolism-related effects with a metabolic chamber. The investigators will test local metabolism with microdialysis during exercise routines, and the investigators will perform fat and muscle biopsies to investigate tissue-related effects. The investigators include experience from a broad-ranging spectrum. The investigators findings might improve understanding mechanisms linking physical exercise and endogenous metabolism. Furthermore, they could influence decision-making regarding non-pharmacological interventions.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index 27-40 kg/m2
* Abdominal obesity (waist circumference >102 cm form men, >88 cm for women)
* Two further diagnostic criteria of metabolic syndrome (ATP III Definition):
* HDL cholesterin <40 mg/dl for men, <50 mg/dl for men
* Triglyceride >150 mg/dl
* Fasting glucose >110 mg/dl
* Blood pressure >135/80 mm Hg
* Less than 2 hours of physical activity per week
* Sinus rhythm

Exclusion Criteria:

* Other relevant metabolic or cardiovascular diseases

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2012-01; Primary Completion 2017-07 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Increase in mitochondria number in skeletal muscle with exercise in hypoxia compared to normoxia | Participants will be followed for the duration of the training program, an expected average of 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Charite University Medicine, ECRC, Berlin, Germany